CLINICAL TRIAL: NCT04897035
Title: A Non-randomized, Open-Label Study to Evaluate the Safety and Effectiveness of Dayspring Active Wearable Compression Technology for Treating Lower Extremity Lymphedema
Brief Title: Study to Evaluate the Safety and Effectiveness of Dayspring for Lower Extremity Lymphedema
Acronym: TIBER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Koya Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KCT 006
Record Dates: First submitted 2021-05-12; First posted 2021-05-21 (Actual); Results first posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2021-05

CONDITIONS: Lymphedema; Lymphedema Lower Extremity; Chronic Venous Insufficiency; Secondary Lymphedema
MeSH Terms: conditions — Lymphedema

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Subjects with Lower Extremity Lymphedema and phlebolymphedema (Experimental): Lower Extremity Lymphedema and phlebolymphedema
  Interventions: Device: Dayspring Active Wearable Compression System

INTERVENTIONS:
Device: Dayspring Active Wearable Compression System — Dayspring Active Wearable Compression System

SUMMARY:
A Non-randomized, Open-Label Study to Evaluate the Safety and Effectiveness of Koya Dayspring Active Wearable Compression Technology for Treating Lower Extremity Lymphedema

ELIGIBILITY:
Inclusion Criteria:

* Males and females ≥ 18 years of age
* Willing to sign the informed consent and deemed capable of following the study protocol
* Subjects must have a diagnosis of primary or secondary unilateral lower extremity edema
* At the time of initial evaluation, individuals must be at least 3 months post surgery, chemotherapy and/or radiation treatment for cancer if applicable

Exclusion Criteria:

* Individuals with a history or presence of an acute systemic disorder or condition that could place the patient at increased risk from sequential compression therapy
* Inability or unwillingness to participate in all aspects of study protocol and/or inability to provide informed consent
* Patients with exam results that would prevent safe and effective use of the study device (cellulitis, open-wounds, healing-wounds, etc.)
* Patients must not have any diagnosed cognitive or physical impairment that would interfere with use of the device
* Diagnosis of lipedema
* Diagnosis of active or recurrent cancer (< 3 months since completion of chemotherapy, radiation therapy or primary surgery for the cancer)
* Diagnosis of Acute infection (in the last four weeks)
* Diagnosis of acute thrombophlebitis (in last 6 months)
* Diagnosis of pulmonary embolism or deep vein thrombosis within the previous 6 months
* Diagnosis of pulmonary edema
* Diagnosis of congestive heart failure (uncontrolled)
* Diagnosis of chronic kidney disease with acute renal failure
* Diagnosis of epilepsy
* Patients with poorly controlled asthma
* Any condition where increased venous and lymphatic return is undesirable
* Women who are pregnant, planning a pregnancy or nursing at study entry
* Participation in any clinical trial of an investigational substance or device during the past 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-07-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - PT works, Los Altos, California
  - Ginger-K Lymphedema & Cancer Center, Morgan Hill, California

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Subjects With Lower Extremity Lymphedema and Phlebolymphedema
Started | 24
Completed | 24
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: No difference - all participants were assigned to the study group
Arm/Group | Subjects With Lower Extremity Lymphedema and Phlebolymphedema
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 63 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 22
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: LYMQOL (LYMphedema Quality of Life) ***All Relevant Time Points Used in the Calculation in the Time Frame (e.g., Baseline and 3 Months).***
Description: The Lymphedema Quality of Life Questionnaire (LYMQOL), a validated disease-specific QoL tool, was also administered at baseline and at month 3. Overall QoL is scored on a single item by the patient on a scale of 1-10. The outcome measure is assessed as a difference or change from baseline LYMQOL at day zero and month 3.
  Higher value is better on the QoL outcome and is more favorable.
Time Frame: 3 months
Population: Higher value is better on the QoL outcome and is more favorable. The difference greater than 0 between baseline and end of study is more favorable
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Subjects With Lower Extremity Lymphedema and Phlebolymphedema
Number analyzed (Participants) | 24
units on a scale | .83 (.02)

2. Primary Outcome: Change in Edema Volume
Description: Change in edema volume is measured as the difference between the edema volume at 3 months and edema volume at baseline. Edema volume is the difference in volume between the affected and unaffected limb. Limb volume measurement is performed by using a calibrated tape measure to measure circumference from the ankle and at 4cm increments to the waist region. Measurements are taken for both lower extremities. Volume is calculated based on cylindrical segment analysis.
  A greater change in edema volume between the two time points is better on reduction of limb volume/swelling.
Time Frame: 3 months
Population: Higher value is better on reduction of limb volume/swelling.
Measure: Mean (Standard Deviation); unit: Mean change in edema volu,e, cm3
Arm/Group | Subjects With Lower Extremity Lymphedema and Phlebolymphedema
Number analyzed (Participants) | 24
Mean change in edema volu,e, cm3 | 427.1 (56)

3. Secondary Outcome: Safety/AEs
Description: As assessed by reported adverse events
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Subjects With Lower Extremity Lymphedema and Phlebolymphedema
Number analyzed (Participants) | 24
Participants | 0

4. Secondary Outcome: Number of Patients Using the Device Every Day for at Least 45 Minutes
Description: Outcome measure will be evaluated based on number of patients that have used the device for the recommended use of 45 minutes per day over the duration of 3 months.
Time Frame: 3 months
Measure: Number; unit: Patients using device every day
Arm/Group | Subjects With Lower Extremity Lymphedema and Phlebolymphedema
Number analyzed (Participants) | 24
Patients using device every day | 24

ADVERSE EVENTS:
Time Frame: 1 year
Description: This study involves a Class II, FDA-cleared medical device used within its cleared indication and standard clinical practice. The device is non-implantable, non-life-sustaining, and non-systemic, with no plausible mechanism by which its use could result in death.
  Study participation does not introduce procedures or conditions associated with mortality risk. Therefore, all-cause mortality is not a relevant safety endpoint, and no participants are considered at risk.
Arm/Group | Subjects With Lower Extremity Lymphedema and Phlebolymphedema
All-Cause Mortality (participants affected / at risk) | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24
Other Adverse Events (participants affected / at risk) | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2021-01-01): https://cdn.clinicaltrials.gov/large-docs/35/NCT04897035/Prot_001.pdf